CLINICAL TRIAL: NCT05275933
Title: Assessing the Efficacy of TCM Capsules Lian Hua Qing Wen Jiao Nang as Adjuvant Treatment in Mild COVID-19 Patients on Home Recovery Program in Singapore: a Randomised, Double-blind, Placebo-controlled Study
Brief Title: Efficacy of TCM Capsules Lian Hua Qing Wen Jiao Nang in Mild COVID-19 Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Singapore Chung Hwa Medical Institution (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCHMI-2021-001
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: A randomised, double-blind, placebo-controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PC+SC (Placebo Comparator): Placebo Control Capsules (PC) are provided in addition to Standard Care medications
  Interventions: Other: Placebo intervention
- LH+SC (Active Comparator): Lian Hua Qing Wen Capsules (LH) are provided in addition to Standard Care medications.
  Interventions: Other: TCM intervention

INTERVENTIONS:
Other: TCM intervention — Lian Hua Qing Wen Capsules (LH) are provided in addition to Standard Care medications which include Symptomatic therapies include Paracetamol, antihistamines (eg. Cetirizine, loratadine or chlorpheniramine) and etc pro re nata (PRN) basis accordingly to the patient's condition.
  Arms: LH+SC
Other: Placebo intervention — Placebo Capsules (PC) are provided in addition to Standard Care medications which include Symptomatic therapies include Paracetamol, antihistamines (eg. Cetirizine, loratadine or chlorpheniramine) and etc pro re nata (PRN) basis accordingly to the patient's condition.
  Arms: PC+SC

SUMMARY:
This research aims to investigate the adjuvant effect of LH in reducing the symptomatic duration of fully vaccinated, mild COVID-19 patients on home recovery program in Singapore. It is aimed to assist policymakers in incorporating clinically proven TCM treatment for mild COVID-19 patients on home recovery program, and establishing a guideline on TCM pandemic treatment protocol which is suitable to be integrated into the healthcare system.

DETAILED DESCRIPTION:
Importance With the emergence of Covid-19 variants and despite having 93% population vaccination rate, the daily number of community cases in Singapore is still surging. Lian Hua Qing Wen Capsules (LH) was reported to have effective inhibitory action on Delta SARS-CoV-2 in-vitro. Due to limited availability and prioritisation of approved anti-viral drugs (Paxlovid) to moderate and severe inpatients, validating Traditional Chinese Medicine (TCM) intervention LH as a good adjuvant treatment for local population on home recovery program is important.

Objectives This research aims to investigate the adjuvant effect of LH in reducing the symptomatic duration of fully vaccinated, mild COVID-19 patients on home recovery program in Singapore. It is aimed to assist policymakers in incorporating clinically proven TCM treatment for mild COVID-19 patients on home recovery program, and establishing a guideline on TCM pandemic treatment protocol which is suitable to be integrated into the healthcare system.

Hypothesis The investigators hypothesize TCM intervention could shorten (1) the time of 8 major clinical symptoms of COVID-19 to no symptoms and (2) lesser days to COVID-19 Antigen Rapid Test (ART) negativity by 1.5 times in mild COVID-19 patients on home recovery program.

Methods 300 eligible participants will be enrolled. Equal number of participants will be randomised and double blinded in the two arms of placebo control and LH, both with standard care. Communication and consultation will be conducted through telecommunication. Primary outcome measures time to no symptoms. Secondary outcomes measure days to ART negativity, symptom severity scores and risk ratio. Exploratory outcomes include days of TCM Excess syndromes (symptoms caused by pathogenic factors) will be collated.

Significance Adjuvant treatment of mild COVID-19 patients can shorten symptomatic duration, slow disease progression, mitigate post-isolation COVID-19 symptoms, and allow isolated individuals to return to the community earlier.

ELIGIBILITY:
Inclusion Criteria:

1. Participants of age 21 to 79 years, all gender and races.
2. Participant provides informed consent prior to initiation of any study procedures.
3. Fully vaccinated (according to latest MOH criteria. Refer to Appendix 1) and qualified for Protocol 2 Primary Care (P2PC) (Appendix 2).
4. Documentation of confirmed active SARS-CoV-2 infection, as determined by PHPC and MOH.
5. Mild COVID-19 experiencing at least one SARS-CoV-2 infection symptom within the first two days of COVID-19 diagnosis including symptoms of mild illness with COVID-19 (based on Questionnaire 6.2) that could include fever, cough, sore throat, malaise, headache, muscle pain, gastrointestinal symptoms, without shortness of breath or dyspnea, with stable vital signs.
6. Agrees to not participate in another clinical trial for the treatment of COVID-19 or SARS-CoV-2 during the study period up until reaching hospitalization or 28 days, whichever is earliest.
7. Agrees to not utilize TCM or other alternative medicine and supplements outside of this study during the 7-day period.
8. Willing to be randomized to LH and PC arm for 7 days and followed up to 28 days.
9. Willing to comply with the study related questionnaires, procedures, and measurements.
10. Willing to not become pregnant during the 7 days of LH ingestion using appropriate accepted methods of contraception. Acceptable methods of contraception include: postmenopausal 1 year of amenorrhea and over 50 years of age; prior tubal ligation or hysterectomy; or barrier contraception using condom or diaphragm plus spermicide.
11. Able to provide the identity of their health care provider or health system clinical care entry information (if any).
12. Able to utilize telephone, WhatsApp apps and/or Online platform (Zoom/ VooV) to comply with the study related questionnaires, procedures, and measurements, established during the recruitment process.
13. Able to speak and communicate in basic English.

Exclusion Criteria:

1. Not fully vaccinated (according to latest MOH criteria. Refer Appendix 1).
2. Patients classified under Protocol 1 according to latest MOH Criteria (Appendix 2) or required hospitalisation (based on PI/Co-I's diagnosis).
3. TCM syndrome of cold deficiencies in spleen and stomach (for example: long-term loose stool), qi and blood debilitation (for example: long-term dizziness).
4. Positive SARS-CoV-2 molecular test in the absence of COVID-19 symptoms from day 1 (Asymptomatic), PCR/ ART test is negative.
5. Moderate, Severe or Critical COVID-19:

   1. Moderate Covid-19: Individuals who show evidence of lower respiratory disease during clinical assessment or imaging and who have an oxygen saturation (SpO2) ≥94% on room air at sea level.
   2. Severe COVID-19: Symptoms suggestive of severe systemic illness with COVID-19, which could include any symptom of moderate illness or shortness of breath at rest, or respiratory distress
   3. Clinical signs indicative of severe systemic illness with COVID-19, respiratory rate ≥ 30 breaths per minute, heart rate ≥ 125 beats per minute, SpO2 ≤ 93% on room air at sea level or respiratory PaO2/FiO2 < 300.
6. Critical COVID-19; Evidence of critical illness, defined by at least one of the following:

   1. Respiratory failure defined based on resource utilization requiring at least one of the following: Endotracheal intubation and mechanical ventilation, oxygen delivered by high flow nasal cannula (heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates > 20 L/min with fraction of delivered oxygen ≥ 0.5), non-invasive positive pressure ventilation, ECMO, or clinical diagnosis of respiratory failure (i.e., clinical need for one of the preceding therapies, but preceding therapies not able to be administered in setting of resource limitation).
   2. Shock (defined by systolic blood pressure < 90 mm Hg, or diastolic blood pressure < 60 mm Hg or requiring vasopressors).
   3. Multi-organ dysfunction/failure.
7. Use of drugs for anti-SARS-CoV-2 treatment including remdesivir, baricitinib, lopinavir/ritonavir fixed dose combination, ribavirin, chloroquine, hydroxychloroquine, and azithromycin, dexamethasone, bamlanivimab, casirivimab plus imdevimab convalescent plasma, or participation in a clinical trial involving any of these drugs whether for treatment or prophylaxis.
8. Participating in a study where co-enrolment is not allowed.
9. Known allergy/sensitivity or any hypersensitivity to components of LH or standard care medication.
10. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
11. Has known prior kidney disease.
12. Has known cirrhosis, acute liver disease or uncontrolled chronic liver disease.
13. Has known narrow angle glaucoma.
14. Has Glucose-6-phosphate dehydrogenase (G6PD) deficiency.
15. On psychiatric medication including Monoamine oxidase inhibitors (MAOIs).
16. If has (a) three or more co-morbidities / chronic conditions even if they are under controlled, or (b) one uncontrolled chronic condition. Chronic diseases include cardiovascular disease (coronary artery disease, heart failure, valvular heart disease), hypertension, diabetes, hyperlipidaemia, chronic lung disease, chronic kidney disease, chronic liver disease, chronic thyroid disease, immunocompromised (HIV or daily users of more than 5 mg/day of prednisone), prior organ transplant, epilepsy.
17. Currently undergoing chemotherapy, radiotherapy, targeted therapy, or immuno-therapy treatment.
18. Fulfils the MOH criteria of at high risk for progressing to severe COVID-19.
19. Women who are currently pregnant or breastfeeding.

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
1.1 Time (Days) to become asymptomatic (the event) for all 8 major COVID-19 symptoms. | up to 7 days after enrolment
  To document the adjuvant effect of LH on Symptom Severity Score within 7 days of enrolment in the PC + standard care and LH + standard care treatment at Day 1 to Day 7 every day.
  8 major Covid-19 symptoms: Stuffy or runny nose, Sore throat, Cough, Low energy or tiredness, Muscle or body aches, Headache, Chills or shivering, Feeling hot or feverish.
  The time (days) to become asymptomatic (the event) is defined as when all the 8 major Covid-19 symptoms meet the criteria of disappearing (score 0) and are stable for at least 24 hours.

SECONDARY OUTCOMES:
2.1 Median Time to COVID-19 ART negativity | up to 7 days after enrolment
  Detection of SARS-CoV-2 viral proteins (antigens) in respiratory tract specimens using a standardised locally approved self-administering Antigen Rapid Test (ART) Kit of the same brand and model daily from Day 1 to Day 7.
  • Time to COVID-19 ART negativity (the event) will be recorded, and are ART negative for the next additional 2 days.
2.2 Symptom Severity Score | up to 7 days and on the 28th day after enrolment
  To investigate symptom recovery and mean reduction score (defined as absolute differences of the overall symptom severity scores from baseline day 1) comparison between 2 arms on days 1-7, 28 specifically.
  * Overall symptom severity score (added together) for the following symptoms will be calculated:
  * Stuffy or runny nose
  * Sore throat
  * Cough
  * Low energy/tiredness
  * Muscle/body aches
  * Headache
  * Chills/shivering
  * Fever/Feeling hot/feverish
  * Sense of smell
  * Sense of taste
    * The lower the score the less intensity the symptoms are. For each symptoms (with specific definitions), 0 point represents no symptoms, 1 point represent mild, 2 point represent moderate and 3 point represents severe.
2.3 Adverse Events | up to 7 days and on the 28th day after enrolment
  To document observed cumulative incidence of adverse events including event that leads to early discontinuation of PC+SC or LH+SC.
  Incidence of serious adverse events including COVID-19 disease worsening requiring medical intervention and/or hospitalization within 28 days will also be recorded and reported.
2.4 Time to become asymptomatic (the event) for the 3 Covid-19 symptoms of interest | up to 7 days after enrolment
  The time (days) to become asymptomatic (the event) for the 3 major Covid-19 symptoms of Stuffy or runny nose, Sore throat and Cough and meet the criteria of disappearing (score 0) and are stable for at least 24 hours.

OTHER OUTCOMES:
3.1 Feasibility of recruitment | 6 months
  To document the feasibility of recruitment through community setting by assessment of the number of positive cases identified per week
3.2 Participation Rate | 6 months
  To document the proportion of patients who agree to participate as measured by enrolment and randomization
3.3 Study agent compliance | up to 28 days after enrolment
  To document the proportion of patients who are compliant taking greater than 90% of the test medicine (including standard care medication) as measured by self-report.
3.4 Symptom monitoring compliance | up to 28 days after enrolment
  To document the proportion of patients who comply with symptom monitoring.
3.5 Discontinuation rate | up to 7 days after enrolment
  To document the proportion of patients who do not complete the clinical trial, including both adverse events related or non-adverse events related.
3.6 TCM Syndrome Differentiation (without pulse taking) | Alternate days up to 7 days, and on the 28th day after enrolment
  To document TCM syndromes and symptoms including TCM tongue observation on alternate days within 7 days of enrolment and on day 28 for post and cross analysis.
  * The lower the score the less intensity the TCM symptoms are. For each TCM symptoms (with specific definitions), 0 represents no symptoms, 1 represent mild, 2 represent moderate and 3 represents severe. TCM scores are not being quantified and used as primary clinical endpoint, together with tongue observation as qualitative measures for diagnosis and record of TCM syndromes.

CONTACTS AND LOCATIONS:
Overall Officials: Sze Tat Ong, MBBS Hons, Principal Investigator — Singapore Chung Hwa Medical Institution
Locations (2):
- Singapore (2):
  - Ubi Family Clinic & Surgery, Singapore
  - Banyan clinic @ jw private limited, Singapore

IPD SHARING:
Plan to Share IPD: Undecided